CLINICAL TRIAL: NCT03865992
Title: Curcumin for Breast Cancer Survivors With Aromatase Inhibitor-Induced Joint Arthropathy - A Randomized, Double-Blinded, Controlled Pilot Study
Brief Title: Curcumin in Reducing Joint Pain in Breast Cancer Survivors With Aromatase Inhibitor-Induced Joint Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18432; NCI-2018-03787 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18432 (Other: City of Hope Medical Center); UG1CA189823 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-03-07 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Joint Pain
Keywords: Breast cancer; curcumin; aromatase inhibitor; joint pain; arthropathy
MeSH Terms: conditions — Breast Neoplasms; Arthralgia; Joint Diseases | interventions — Curcumin; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (nanoemulsion curcumin) (Experimental): Patients receives nanoemulsion curcumin orally (PO) twice daily (BID) for up to 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Curcumin; Other: Nanoemulsion; Other: Quality-of-Life Assessment; Behavioral: Questionnaire
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for up to 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — Given capsules for oral administration
  Other Names: C.I. 75300; C.I. Natural Yellow 3; Diferuloylmethane; Turmeric Yellow; (E,E)-1,7-Bis(4-hydroxy-3-methoxyphenyl)-1,6-heptadiene-3,5-dione, 32982, 458-37-7
  Arms: Arm I (nanoemulsion curcumin)
Other: Placebo — Given capsules for oral administration
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Nanoemulsion — Given nanoemulsion curcumin PO
  Arms: Arm I (nanoemulsion curcumin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment,
  Arms: Arm I (nanoemulsion curcumin)
Behavioral: Questionnaire — Ancillary studies
  Other Names: Questionnaires
  Arms: Arm I (nanoemulsion curcumin)

SUMMARY:
This phase I trial studies how well curcumin works in reducing joint pain in patients who are breast cancer survivors and have joint disease caused by treatment with aromatase inhibitors. Curcumin is an ingredient of turmeric, a plant in the ginger family, which is commonly used in curries and South Asian and Middle Eastern cooking, and may decrease joint pain in patients with arthritis from other conditions (such as osteoarthritis and rheumatoid arthritis).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of using Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) scores to detect changes in AI-induced symptoms and well-being in postmenopausal women with breast cancer at 3 months of nanoemulsion curcumin (NEC) vs placebo

SECONDARY OBJECTIVES:

I. To evaluate Disabilities of the Arm, Shoulder and Hand (DASH), Brief Pain Inventory, and Geriatric Assessment as secondary tools for monitoring AI-induced symptoms and well-being II. To evaluate adherence to a regimen of NEC vs placebo by postmenopausal women experiencing joint arthropathy induced by aromatase inhibitor therapy III. To obtain preliminary data regarding function in women with AI induced arthropathy (IA) by monitoring grip strength at 0 and 3 months of NEC versus placebo IV. To conduct exploratory analyses of blood based biomarkers in postmenopausal women with AI-induced arthropathy taking NEC vs placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nanoemulsion curcumin orally (PO) twice daily (BID) for up to 3 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO BID for up to 3 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed primary invasive adenocarcinoma of the breast, stages I-IIIA
* Estrogen-receptor positive (ER+) and/or progesterone-receptor positive (PR+) breast cancer
* Completion of definitive surgery with mastectomy or breast conserving therapy
* Postmenopausal (no menses >= 12 months) or on ovarian suppression in order to take AIs
* Currently taking an Food and Drug Administration (FDA) approved third-generation aromatase inhibitor (e.g., anastrozole [Arimidex], letrozole [Femara], or exemestane [Aromasin]) for >= 90 days prior to registration with plans to continue for >= 90 days after registration
* Clinical symptoms of joint pain for at least 3 months prior to study entry that started or increased with AI therapy with Brief Pain Inventory (BPI) Worst Pain score >= 4 (verbal response to BPI question 3 regarding the worst pain in the past 24 hours as 0 "no pain" to 10 "pain as bad as you can imagine")

Exclusion Criteria:

* Prior malignancy =< 5 years except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, ductal carcinoma in situ of the breast or adequately treated stage I or II cancer from which the patient is currently in complete remission
* History of a bleeding tendency or current use of coumadin or other anticoagulants
* Current or previous history of anemia
* Current autoimmune, liver, hematopoietic, cardiac, or renal disease
* Current viral, bacterial, atypical or fungal infections of any organ system
* Concurrent use of immunosuppressant medications
* Concurrent use of medications known to inhibit or induce hepatic enzyme CYP 3A4 (e.g. ketoconazole, macrolide antibiotics, barbiturates)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Bone fracture or surgery of the affected joints, within 180 days of study entry
* Medical therapy, alternative therapy, or physical therapy for joint pain/stiffness =< 30 days of study entry
* Intra-articular steroids =< 90 days of study entry or oral/intramuscular corticosteroids < 30 days of entry
* Use of analgesics (e.g., opiates, tramadol with the exception of nonsteroidal anti-inflammatory drugs [NSAIDs] and acetaminophen) within 14 days prior to registration, or at any time during the 3-month study period
* Chronic use of any herbal or dietary supplement containing curcumin or curcuminoids =< 3 months of study entry or any other supplements that might interact with NEC (e.g. St. John's Wort)
* Known sensitivity or allergy to turmeric spices or curry

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Changes in aromatase inhibitor-induced symptoms and overall wellbeing in postmenopausal women on aromatase inhibitor therapy | Up to 3 months
  The study will assess the feasibility of using the Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) to detect changes in aromatase inhibitor (AI)-induced symptoms and well-being in postmenopausal women with breast cancer randomized to 3 months of nanoemulsion curcumin (NEC) versus (vs) placebo capsules.
Change in Brief Pain Inventory (BPI) pain score | Baseline up to 3 months
  The scores obtained from the Disabilities of the Arm, Shoulder and Hand (DASH) and BPI, and FACT-ES assessments will be plotted over time for each arm. The agreement between these instruments will be evaluated using Altman and Bland plot after proper data transformation.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post study-drug assessment
  Adverse events will be characterized using the descriptions and grading scales found in the most recent version of the Common Terminology Criteria for Adverse Events version 5.0.
Change in FACT-ES score | Baseline up to 3 months
  The scores obtained from the BPI, DASH, and FACT-ES assessments will be plotted over time for each arm. The agreement between these instruments will be evaluated using Altman and Bland plot after proper data transformation
Change in DASH score | Baseline up to 3 months
  The scores obtained from the BPI, DASH, and FACT-ES assessments will be plotted over time for each arm. The agreement between these instruments will be evaluated using Altman and Bland plot after proper data transformation.

OTHER OUTCOMES:
Joint symptoms occurrence | Up to 3 months
  The study will use logistic regression models to compare the occurrence of moderate to severe joint symptoms during the 3 month period between the two study groups, with potential covariates including geriatric assessment (GA), age, body mass index, baseline pain scores (0 month), prior chemotherapy e.g. taxanes, time to menopause/ovarian suppression. Summary statistics will be generated using the data obtained from the T0 and T3 study visits where grip strength dynamometry completed. Temporal as well as other relevant correlations between the data and the validated assessment scores will be determined.
Blood based biomarker analysis | Up to 3 months
  The study will explore the relationship between specific inflammatory blood markers, grip strength, and the joint symptoms evaluated by the patient reported outcome measures. The relationship between plasma curcumin and these measures will also be evaluated. Scatter plots and correlation coefficients (either Pearson or Spearman) will be used to summarize their pair wise relation. The differences between the treatment and placebo in terms of these measures will also be reported using numerical summaries and graphic plots.
Adherence rates | Up to 3 months
  Adherence rates will be examined using pill counts each month and patient recorded daily logs. Plasma curcumin will be compared to daily logs and pill count data as another potential measure of adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Yee, MD, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope South Pasadena, South Pasadena, California
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Lustberg M, Fan-Havard P, Wong FL, Hill K, Phelps MA, Herrera KW, Tsai NC, Synold T, Feng Y, Kalu C, Sedrak MS, Yee LD. Randomized placebo-controlled, double-blind clinical trial of nanoemulsion curcumin in women with aromatase inhibitor-induced arthropathy: an Alliance/NCORP pilot trial. Breast Cancer Res Treat. 2024 May;205(1):61-73. doi: 10.1007/s10549-023-07223-4. Epub 2024 Jan 27. PMID 38280052